CLINICAL TRIAL: NCT03223532
Title: A Prospective, Randomized, Open Label Trial Comparing PrePex™ Day 7 Foreskin Removal Procedure (FRP) to a PrePex Day 0 FRP of Male Circumcision in Resource Limited Settings
Brief Title: Randomized Trial Comparing PrePex Day 7 Foreskin Removal Procedure (FRP) to a Day 0 PrePex FRP .
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nyanza Reproductive Health Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VMMC005
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Male Circumcision

STUDY DESIGN:
Intervention Model Description: A Prospective, Randomized, Open Label Trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrePex Day 7 FRP (Active Comparator): Standard PrePex procedure, 1 week after device placement foreskin and device are removed.
  *Subjects must be adequately vaccinated, or willing to be vaccinated, against Tetanus based on appropriate national guidance for male circumcision
  Interventions: Device: PrePex Day 7 FRP
- PrePex Day 0 FRP (Experimental): On the day of device placement the foreskin is removed, the device is removed 1 week later.
  Interventions: Device: PrePex Day 0 FRP

INTERVENTIONS:
Device: PrePex Day 7 FRP — Standard PrePex procedure, foreskin and device are removed 1 week after device application.
  Arms: PrePex Day 7 FRP
Device: PrePex Day 0 FRP — Removal of the foreskin shortly after device application, the device is removed 1 week later
  Arms: PrePex Day 0 FRP

SUMMARY:
A Prospective, Randomized, Open Label Trial Comparing PrePex™ Day 7 (FRP) to a PrePex Day 0 FRP of Male Circumcision in Resource Limited Settings.

DETAILED DESCRIPTION:
Study Objectives:

To compare the safety and acceptability of PrePex Day 7 Foreskin Removal Procedure (FRP) (herein: PrePex) versus PrePex Day0 FRP

Planned Subjects Population:

One hundred and fifty (150) subjects scheduled for voluntary medical male circumcision. The subjects will be randomly divided into two unbalanced study arms (2:1), Day0 FRP arm which will include hundred (100) subjects and PrePex arm which will include fifty (50) subjects.

Study duration per subject will be up to 7 weeks and will include a total of 9 visits.

Study Site: University of Nairobi, Illinois, and Manatoba (UNIM) Research and Training Centre, Kisumu, Kenya

ELIGIBILITY:
Inclusion Criteria:

* Ages - 13 to 49 years
* Uncircumcised
* Adequately vaccinated, or willing to be vaccinated, against Tetanus based on appropriate national guidance for male circumcision
* Willing to be circumcised
* Legal guardian consent to the procedure for ages 13-18 years
* Agrees to be circumcised by any of the study methods, Day0 FRP or Day7 FRP as will be determined randomly
* Able to understand the study procedures and requirements
* Agrees to abstain from sexual intercourse for 8 weeks after circumcision
* Agrees to abstain from masturbation for at least 2 weeks after Removal
* Agrees to return to the health care facility for follow-up visits (or as instructed) after his circumcision for a period of 6 weeks post removal (7 weeks total)
* Subject able to comprehend and freely give informed consent for participation in this study and is considered by the investigator to have good compliance for the study

Exclusion Criteria:

* Legal guardian withholds consent for ages 13-18 years
* Active genital infection, anatomic abnormality or other condition, which in the opinion of the investigator prevents the subject from undergoing a circumcision
* Subject with the following diseases/conditions: phimosis, paraphimosis, adhesions, warts under the prepuce, torn or tight frenulum, narrow prepuce, hypospadias, epispadias
* Known bleeding / coagulation abnormality, uncontrolled diabetes
* Subject that to the opinion of the investigator is not a good candidate
* Subject does not agree to anonymous video and photographs of the procedure and follow up visits.

Ages: 13 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Uncircumcised males willing to undergo the non-surgical PrePex male circumcision procedure
Enrollment: 152 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2017-10-14 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events related to the Day 0 FRP | 8 weeks
  Assessing the safety of PrePex Day 0 FRP compared to the standard Day 7 FRP, by means of the following parameter: Incidence of Serious Adverse Events.

SECONDARY OUTCOMES:
Acceptability of PrePex Day 0 FRP | 8 weeks
  Evaluating the PrePex Day 0 FRP acceptability to subjects and health care providers compared to the standard Day 7 FRP, by means of the following parameters:
  1. Evaluation of pain by the following parameters: Subject's subjective pain, tingling and discomfort
  2. Odour assessment while device is in situ by means of questionnaires on follow up visit 3 and on removal visit day.
  3. Subjects / health care providers satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Fredrick Otieno, M.D., Principal Investigator — Nyanza Reproductive Health Society
Locations (1):
- Nyanza Reproductive Health Society, Kisumu, Nyanza, Kenya

IPD SHARING:
Plan to Share IPD: No